CLINICAL TRIAL: NCT05295264
Title: Active Pregnancy. Mental and Emotional Health Care to Pregnant Woman During and After COVID-19
Brief Title: Active Pregnancy. Mental and Emotional Health Care to Pregnant Woman During and After Coronavirus (COVID-19)
Acronym: GESTACTIVE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Politecnica de Madrid (Other)
Collaborators: Hospital Severo Ochoa (Other); Puerta de Hierro University Hospital (Other); Hospital Universitario de Torrejón,Madrid (Other); Hospital Clinic of Barcelona (Other); Hospital Vall d'Hebron (Other); Clinica Zuatzu (Unknown)
Responsible Party: Principal Investigator, Rubén Barakat Carballo, Doctor, Universidad Politecnica de Madrid
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Gestactive2022
Record Dates: First submitted 2022-03-24; First posted 2022-03-25 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Mental Health Wellness; Emotional Problem
Keywords: pregnancy; exercise; lifestyle; physical activity; fetal-maternal health
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): The design of the physical exercise program will be supported by the Canadian and Spanish Guidelines for exercise throughout pregnancy and published by Barakat model.
  Frequency: The program will consist of three weekly sessions. The duration of every session will be 55-60 minutes. The intensity of the workload will be 55-60% of the maximum maternal Heart Rate, and controlled by Polar monitor (FT60). Likewise, once a week, the Borg Scale of Perceived Effort will be administered to participants, in order to have a more reliable assessment of the intensity of the activities, 12-14 (moderate; out of a 20 point scale) will be the level used.
  The minimum adherence required for the participants will be 80% of the total sessions (approximately 80 sessions).
  Interventions: Other: Moderate exercise program
- Control group (No Intervention): Women randomly assigned to the control group (CG) received general advice from their health care provider about the positive effects of physical activity. Participants in the CG had their usual visits with health care providers during pregnancy, which were equal to the exercise group. Women were not discouraged from exercising on their own. However, women in the CG were asked about their exercise once each trimester using a "Decision Algorithm" (by telephone).

INTERVENTIONS:
Other: Moderate exercise program — Exercise program All sessions will begin with a warm-up of 7-8 minutes composed of mild movements and joint mobility of upper and lower limbs exercises. Then a central part of 35-40 minutes, four types of activities will be included (aerobic work, muscle strengthening, coordination/balance tasks, pelvic floor exercises), finally a section of flexibility, relaxation, and final talk (comments and sharing) will be performed (12-15 minutes).
  Healthy lifestyle advise This intervention consists of providing guidelines and videos with advice on healthy habits throughout the pregnancy process. This type of content will be related to daily physical activity, food recommendations, and fundamental exercises to perform during pregnancy.
  Arms: Exercise group

SUMMARY:
The complex process of pregnancy and childbirth can determine the future health of mother and child. It is the only vital process that involves the modification of practically all of a woman's body systems in order to sustain fetal life. In this sense, it is essential to ensure adequate functioning of all maternal physiological, mental and emotional mechanisms that facilitate fetal growth and development. Complications in any of these health domains and functions may contribute to pathologies and complications that have a detrimental impact on maternal and newborn health.

Pregnancy could be a vulnerable period for women, especially regarding mental and emotional illnesses, which are more likely to manifest during this time compared to other periods of their life. In this sense, a high prevalence of prenatal stress, anxiety and depression exists, which are associated with downstream newborn complications as well.

Depressive symptoms such as sadness, decreased interest in everyday activities, reduced energy and concentration are generated by the aforementioned gestational lability, these symptoms would appear (mostly) at the beginning of the pregnancy. Feelings of being overwhelmed, uneasiness, threat or imminent danger, uncertainty, difficulty in making decisions, obsessive thoughts could be caused by prenatal anxiety.

According to scientific literature, the consequences of mental and emotional disturbances during pregnancy go beyond the gestational period and affect mother, fetus, newborn, and even child development, including complications such as preterm delivery, prolonged and more instrumental labor, low birth weight, pre-term birth, infant's physical and cognitive developmental delay, and the poor mother-infant relationship.

DETAILED DESCRIPTION:
COVID-19. Risks associated with an inactive pregnancy:

The impact of COVID-19 has generated a global crisis never before experienced, which affects physiological, emotional, mental, and social factors for all population groups, including those who are pregnant with important related risks.

The complications associated with confinement (no group support, reduced mobility, the distance between people, etc.), significantly affects the lifestyle of pregnant individuals and potentially remove one of the basic recommendations established by the international scientific community: a physically active lifestyle.

Scientific evidence confirms that engaging in an unhealthy lifestyle during pregnancy, including inactivity, enhances the risk of chronic disease for both mother and fetus. In fact, the growing epidemic of sedentary behavior affects pregnancy and childbirth with adverse pre, peri, and postnatal outcomes. Unfortunately, the situation caused by COVID-19 could further exacerbate sedentary behavior and its associated complications for pregnant women.

Current Status:

Before the COVID-19 pandemic, the range of prenatal mental and emotional alterations was close to 15-30%, the prevalence being particularly high in low- and middle-income countries. However, the new social and economic situation generated by the COVID-19 pandemic has raised these values significantly, in this sense 37% reported clinically relevant symptoms of depression and 57% of pregnant women experienced symptoms of anxiety.

This means that the pandemic has negatively affected the mental and emotional health of pregnant women, and consequently of future generations. It is necessary (urgent) to intervene right now with preventive policies and alternatives.

The difficulty and associated (maternal/fetal) risks of pharmacological treatment of mental and emotional illnesses during pregnancy, requires the scientific search for new alternatives, especially aimed at the prevention of these pathologies.

There are important lifestyle recommendations promoted by the scientific community about establishing elements that ensure a healthy pregnancy. However, a small percentage of pregnant women meet global healthy lifestyle guidelines. In fact, the scientific literature reports an increase of perinatal disorders, for example, a high percentage of women continue to gain excessive weight during pregnancy in spite of mentioned health recommendations, and this in turn also increases the risk for other complications.

There are no official estimates of healthcare costs that these complications generate but obviously, we speculate significant amounts.

Worldwide, 80% of pregnant women or (or maybe more) don´t achieve the minimum weekly amount of 150 minutes of moderate physical activity intensity. In Spain, this inactivity is similar to other countries, with approximately 19.7% of women achieving the American College of Obstetricians and Gynecologists (ACOG) recommendations to be active weekly during pregnancy.

Physical exercise as a preventive factor:

Given this complex problem, it is necessary (urgent) to find non-invasive prevention mechanisms to benefit the wellbeing of the mother and her child, taking into account that pregnancy predisposes the woman to a significant change in lifestyle.

As substantiated by scientific evidence, physical exercise during pregnancy does not cause adverse effects on the mother and fetus. Indeed, physical exercise during pregnancy may prevent chronic disease risk in the mother and fetus.

Although the scientific literature is not entirely conclusive, many studies show the positive influence of a physical activity program during pregnancy on maternal mental and emotional status (even with better benefits if it´s supervised); this could be a good approach to maintain healthy mental wellbeing.

GESTACTIVE will examine the effects of a supervised moderate exercise program during pregnancy as a preventive tool for mental and emotional distress, as well as associated complications. The results of this proposal will contribute to the improvement of the quality of life of pregnant women and thus the promotion of health of future generations.

Hypothesis Aerobic, moderate, and supervised exercise during pregnancy can be an efficient element of the prevention of mental and emotional alterations that the situation generated by COVID-19 causes to the healthy pregnant population and their children.

Objective Examine the influence of a supervised aerobic exercise program during pregnancy, in non-face-to-face and face-to-face ways, on the prevention of maternal mental and emotional health, fetal, newborn, and infant outcomes during the pandemic state and in the near future.

Material and Methods:

- Study design. A randomized clinical trial (RCT) will be carried out, not masked with healthy pregnant women, giving rise to two study groups: exercise group (EG), pregnant women participating in a regular program of supervised physical exercise and control group ( CG), pregnant women who receive normal obstetric monitoring of their pregnancy, including recommendations regarding dietary-nutritional factors, as well as the benefits of an active pregnancy. All selected pregnant women will sign an Informed Consent before participating in the study.

Women randomly assigned to the CG received general advice from their health care provider about the positive effects of physical activity. Participants in the CG had their usual visits with health care providers during pregnancy, which were equal to the exercise group. Women were not discouraged from exercising on their own. However, women in the CG were asked about their exercise once each trimester using a "Decision Algorithm" (by telephone).

Intervention

General characteristics of the physical exercise program:

* The minimum adherence required will be 80% of the total sessions.
* Onset: gestational week 9-11, immediately after the first prenatal ultrasound, in order to rule out Obstetric Contraindications for physical exercise.
* End: gestational week 38-39.
* Frequency: 3 weekly sessions, various possibilities will be offered at different times from which the pregnant woman can choose, in order to promote work and family conciliation.

Basic Considerations:

a, All the activities carried out will be aerobic.

b. Avoid working positions in which areas normally overloaded by pregnancy are further affected.

c. The work corresponding to flexibility will be carried out always bearing in mind that these are pregnant women, this forces us once again not to include forced operating positions in the exercises or to excessively maintain the stretching times in each area.

d. An adequate fluid intake will be maintained before and after the activity.

e. Also as a general rule and to eliminate potential risks, the following will be avoided:

* Activities that include the Valsalva maneuver.
* High ambient temperatures or very humid environments in order to avoid hyperthermia (body temperature higher than 38º C).
* Sudden movements.
* Positions of extreme muscular tension.

Structure:

All sessions will begin with a warm-up of 7-8 minutes composed of mild movements and joint mobility of upper and lower limbs exercises. Then a central part of 35-40 minutes, four types of activities will be included (aerobic work, muscle strengthening, coordination/balance tasks, pelvic floor exercises), finally a section of flexibility, relaxation and final talk (comments and sharing) will be performed (12-15 minutes).

Below we offer a greater detail of each part:

I. Warm-up-General activation. Displacements varied without impact activities (avoiding jumps, falls). Mild work of mobility of the main joints.

II. Aerobic section. Exercise to increase intensity up to moderate activities, play with sports equipment (balls, ropes, pikes), or choreographies of different musical styles.

III. Muscle strengthening, general toning exercises of the whole body: lower part (calf, quadriceps, hamstrings, adductors, abductors), upper part (abdominal, pectoral, shoulders, paravertebral musculature). Also exercises for the most weakened and needy muscle groups during pregnancy, the aim is to avoid muscular decompensation.

IV. Coordination and balance exercises: simple tasks of eye-hand and eye-foot coordination with sports equipment, as well as body axis balance exercises.

V. Strengthening the pelvic floor muscles, Kegel exercises will be applied and is basically composed of contractions (slow and fast) of the different structures of the pelvic floor musculature.

VI. Relaxing section during 7-8 minutes, aiming to gradually lower the intensity of work with flexibility-stretching and relaxation exercises.

VII. Final Talk. This part is intended for pregnant women to express clearly and openly the sensations and perceptions experienced during the session. The reflection of each participant on the effect of physical practice is sought, not only in the physical or physiological aspect but also in the psychic and emotional section. The exchange of impressions between the pregnant women enhances the role of a correctly designed and conducted physical exercise program, as a social mobile of maintenance and improvement of the quality of life of the pregnant woman.

ELIGIBILITY:
Inclusion Criteria:

- Pregnant women fulfilling the following criteria: >18 years old, singleton pregnancies and planning management and delivery at the research hospitals, and also do not participate in any other program of supervised physical exercise.

Exclusion Criteria:

Women with absolute contraindications. Women with relative contraindications need permission from obstetric care providers prior to participation:

Absolute contraindications to exercise:

* Ruptured membranes.
* Premature labor.
* Unexplained persistent vaginal bleeding.
* Placenta praevia after 28 weeks gestation.
* Pre-eclampsia.
* Incompetent cervix.
* Intrauterine growth restriction.
* High-order multiple pregnancies (eg, triplets).
* Uncontrolled type I diabetes.
* Uncontrolled hypertension.
* Uncontrolled thyroid disease.
* Other serious cardiovascular, respiratory, or systemic disorders.

Relative contraindications to exercise:

* Recurrent pregnancy loss.
* Gestational hypertension.
* A history of spontaneous preterm birth.
* Mild/moderate cardiovascular or respiratory disease.
* Symptomatic anemia.
* Malnutrition.
* Eating disorder.
* Twin pregnancy after the 28th week.
* Other significant medical conditions.

Women in the CG were asked about their exercise once each trimester using a "Decision Algorithm" and those who are excessively actives were excluded.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 500 (Estimated)
Dates: Start 2022-03-17 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Prenatal depression (CES-D) | 9 months
  analyze with a questionnaire the variability during pregnancy (Likert scale 0-3)
Prenatal anxiety, State-Trait Anxiety Inventory (STAI) | 9 months
  analyze with a questionnaire the value and its interrelationship with physical exercise patterns (Likert scale 0-3)
Prenatal stress, Perceived Stress Scale (PSS) | 9 months
  analyze with a questionnaire the value and its interrelationship with physical exercise patterns(Likert scale 0-3)
Postnatal depression, Edinburgh Postnatal Depression Scale (EPDS). | 6 months
  analyze with a questionnaire the value and its interrelationship with physical exercise during pregnancy(Likert scale 0-5)
Postnatal anxiety, State-Trait Anxiety Inventory (STAI) | 6 months
  analyze with a questionnaire the value and its interrelationship with physical exercise patterns (Likert scale 0-3)
Postnatal stress, PSS (Perceived Stress Scale) | 6 months
  analyze with a questionnaire the value and its interrelationship with physical exercise patterns(Likert scale 0-5; higher scores mean a worse outcome)

SECONDARY OUTCOMES:
Maternal weight gain | 9 months
  analyze the increase during pregnancy
Blood pressure | 9 months
  analyze how it varies during pregnancy
O'Sullivan test (OGTT) | 1 month
  analyze the value and its interrelationship with physical exercise patterns
Urinary Incontinence Questionnaire (ICIQ-SF) | 9 months
  analyze with a questionnaire the value and its interrelationship with physical exercise patterns (different measures in the questionnaire)(Likert scale 0-5; higher scores mean a worse outcome)
Behavior of Fetal Heart Rate | 3 months
  analyze variability during pregnancy
Gestational age | 9 months
  analyze the value and its interrelationship with physical exercise patterns
Type of delivery (Vaginal, instrumental or cesarean) | 1 month
  analyze whether women have had a vaginal, instrumental, or cesarean delivery and its interrelationship with physical exercise patterns
Duration of labor | 1 month
  analyze the value and its interrelationship with physical exercise patterns
Birthweight | 1 month
  analyze the value and its interrelationship with physical exercise patterns
Child's weight | 24 months
  analyze the value and its interrelationship with physical exercise patterns during pregnancy
Child's height | 24 months
  analyze the value and its interrelationship with physical exercise patterns during pregnancy
Mental assessment of the child (depression questionnaire adapted to childhood) | 24 months
  analyze the value and its interrelationship with physical exercise patterns during pregnancy (Likert scale 0-3)
Psychomotor behavior of the child | 24 months
  analyze some variables (sitting, crawling, standing, walking, holding objects...) and its relationship with maternal exercise
Maternal pains during pregnancy (headache, back pain, pelvic pain, paravertebral, scapular, etc.) | 9 months
  analyze the value and its interrelationship with physical exercise patterns
Fetal growth and development | 9 months
  analyze the value and its interrelationship with physical exercise patterns
Delivery tears | 1 month
  analyze the value and its interrelationship with physical exercise patterns
Performing episiotomy during childbirth | 1 month
  analyze the appearance (descriptive: yes/no) and its interrelationship with physical exercise patterns
Apgar Score | 1 month
  analyze the value and its interrelationship with physical exercise patterns (1 to 10)
Birth length | 1 month
  analyze the value and its interrelationship with physical exercise patterns
Head circumference | 1 month
  analyze the value and its interrelationship with physical exercise patterns
Landau reflexes test | 1 month
  analyze the value and its interrelationship with physical exercise pattern
Neonatal intensive care unit (NICU) | 1 month
  analyze the number of admissions and its interrelationship with physical exercise patterns
Postpartum recovery of pre-pregnancy weight | 12 months
  analyze how it varies during postpartum period
Umbilical cord Ph | 1 month
  analyze the value and its interrelationship with physical exercise patterns
Fetal development | 9 months, once a trimester
  analyze variables (estimated fetal weight, Fetal cardiac function, fetal measures, uterine arteries...) by ultrasound
Carotid intima-media thickness (CIMT) | 9 months
  Measurement of carotid intima-media thickness (CIMT) with B-mode ultrasound is a noninvasive, sensitive, and reproducible technique for identifying and quantifying subclinical vascular disease and for evaluating cardiovascular disease (CVD) risk.
Maternal sleep habits | 9 months
  analyze with Pittsburgh´s sleep quality index (Likert scale 0-5; higher scores mean a worse outcome)
Maternal body self-perception | 9 months
  analyze using Ben-Toby Walker Body Attitude Questionnaire (Likert scale 0-5; higher scores mean a worse outcome)
Newborn sleep habits | 24 months
  analyze using Brief Infant Sleep Questionnaire (Likert scale 0-5; higher scores mean a worse outcome)
Perception of health status - Short Form 36 health scale | 9 months
  analyze the value and its interrelationship with physical exercise patterns (Likert scale 0-5; higher scores mean a better outcome)
Placental angiogenic factors | measured at 24-25 weeks and at 34-35 weeks
  placental growth factor (PIGF)
Placental angiogenic factors | measured at 24-25 weeks and at 34-35 weeks
  soluble fms-like tyrosinekinase-1 (sFlt1)
Lipidic profile | measured at 24-25 weeks and at 34-35 weeks
  ( Total Cholesterol, LDL-Cholesterol, HDL- Cholesterol, Tryglicerids)

OTHER OUTCOMES:
Recovery of pelvic floor muscles ultrasound | 6 months
  analyze the diameter and thickness of muscles in the perineal area and their interrelationship with physical exercise patterns
Maternal habits of physical activity - Pregnancy Physical Activity Questionnaire (PPAQ) | 12 months
  analyze with a questionnaire how it varies during and after pregnancy
Pregestational maternal patterns | 9 months
  analyze sociodemographic and behavioral habits like (smoking, alcoholism, previous illness, COVID-19, parity, occupation, previous miscarriage...)
Coronavirus disease | 9 months
  analyze the coronavirus condition during pregnancy and its interrelationship with other variables

CONTACTS AND LOCATIONS:
Overall Officials: Rubén Barakat, PhD, Study Director — Universidad Politécnica de Madrid (UPM)
Locations (1):
- Facultad de Ciencias de la Actividad Física y el Deporte - INEF, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khaire A, Wadhwani N, Madiwale S, Joshi S. Maternal fats and pregnancy complications: Implications for long-term health. Prostaglandins Leukot Essent Fatty Acids. 2020 Jun;157:102098. doi: 10.1016/j.plefa.2020.102098. Epub 2020 Apr 21. PMID 32380367
- [Background] Abbasi H, Puusepp-Benazzouz H. Pregnancy Stress, Anxiety, and Depression Sequela on Neonatal Brain Development. JAMA Pediatr. 2020 Sep 1;174(9):908. doi: 10.1001/jamapediatrics.2020.1073. No abstract available. PMID 32568372
- [Background] Wenzel ES, Gibbons RD, O'Hara MW, Duffecy J, Maki PM. Depression and anxiety symptoms across pregnancy and the postpartum in low-income Black and Latina women. Arch Womens Ment Health. 2021 Dec;24(6):979-986. doi: 10.1007/s00737-021-01139-y. Epub 2021 May 10. PMID 33970310
- [Background] Li H, Bowen A, Bowen R, Muhajarine N, Balbuena L. Mood instability, depression, and anxiety in pregnancy and adverse neonatal outcomes. BMC Pregnancy Childbirth. 2021 Aug 25;21(1):583. doi: 10.1186/s12884-021-04021-y. PMID 34429072
- [Background] Graham RM, Jiang L, McCorkle G, Bellando BJ, Sorensen ST, Glasier CM, Ramakrishnaiah RH, Rowell AC, Coker JL, Ou X. Maternal Anxiety and Depression during Late Pregnancy and Newborn Brain White Matter Development. AJNR Am J Neuroradiol. 2020 Oct;41(10):1908-1915. doi: 10.3174/ajnr.A6759. Epub 2020 Sep 10. PMID 32912873
- [Background] Hunter SK, Freedman R, Law AJ, Christians U, Holzman JBW, Johnson Z, Hoffman MC. Maternal corticosteroids and depression during gestation and decreased fetal heart rate variability. Neuroreport. 2021 Oct 6;32(14):1170-1174. doi: 10.1097/WNR.0000000000001711. PMID 34284445
- [Background] Ullah R, Hasan TN, Rahman MU, Naqvi SS, Sharif N, Ahmad I, Ullah B, Khan I, Ammad M, Arshad N. Coronavirus Family: Responsible Agents for Stress, Depression, and Anxiety during Pregnancy. Psychiatr Danub. 2021 Fall;33(3):425-426. No abstract available. PMID 34795194
- [Background] Bivia-Roig G, La Rosa VL, Gomez-Tebar M, Serrano-Raya L, Amer-Cuenca JJ, Caruso S, Commodari E, Barrasa-Shaw A, Lison JF. Analysis of the Impact of the Confinement Resulting from COVID-19 on the Lifestyle and Psychological Wellbeing of Spanish Pregnant Women: An Internet-Based Cross-Sectional Survey. Int J Environ Res Public Health. 2020 Aug 15;17(16):5933. doi: 10.3390/ijerph17165933. PMID 32824191
- [Background] Mottola MF, Davenport MH, Ruchat SM, Davies GA, Poitras VJ, Gray CE, Jaramillo Garcia A, Barrowman N, Adamo KB, Duggan M, Barakat R, Chilibeck P, Fleming K, Forte M, Korolnek J, Nagpal T, Slater LG, Stirling D, Zehr L. 2019 Canadian guideline for physical activity throughout pregnancy. Br J Sports Med. 2018 Nov;52(21):1339-1346. doi: 10.1136/bjsports-2018-100056. PMID 30337460
- [Background] Physical Activity and Exercise During Pregnancy and the Postpartum Period: ACOG Committee Opinion, Number 804. Obstet Gynecol. 2020 Apr;135(4):e178-e188. doi: 10.1097/AOG.0000000000003772. PMID 32217980
- [Background] Meander L, Lindqvist M, Mogren I, Sandlund J, West CE, Domellof M. Physical activity and sedentary time during pregnancy and associations with maternal and fetal health outcomes: an epidemiological study. BMC Pregnancy Childbirth. 2021 Feb 27;21(1):166. doi: 10.1186/s12884-021-03627-6. PMID 33639879
- [Background] Jones MA, Catov JM, Jeyabalan A, Whitaker KM, Barone Gibbs B. Sedentary behaviour and physical activity across pregnancy and birth outcomes. Paediatr Perinat Epidemiol. 2021 May;35(3):341-349. doi: 10.1111/ppe.12731. Epub 2020 Oct 30. PMID 33124060
- [Background] Atkinson L, De Vivo M, Hayes L, Hesketh KR, Mills H, Newham JJ, Olander EK, Smith DM. Encouraging Physical Activity during and after Pregnancy in the COVID-19 Era, and beyond. Int J Environ Res Public Health. 2020 Oct 7;17(19):7304. doi: 10.3390/ijerph17197304. PMID 33036326
- [Background] Dadi AF, Miller ER, Bisetegn TA, Mwanri L. Global burden of antenatal depression and its association with adverse birth outcomes: an umbrella review. BMC Public Health. 2020 Feb 4;20(1):173. doi: 10.1186/s12889-020-8293-9. PMID 32019560
- [Background] Lebel C, MacKinnon A, Bagshawe M, Tomfohr-Madsen L, Giesbrecht G. Elevated depression and anxiety symptoms among pregnant individuals during the COVID-19 pandemic. J Affect Disord. 2020 Dec 1;277:5-13. doi: 10.1016/j.jad.2020.07.126. Epub 2020 Aug 1. PMID 32777604
- [Background] Kolding L, Ehrenstein V, Pedersen L, Sandager P, Petersen OB, Uldbjerg N, Pedersen LH. Obstetric care for women that use antidepressants in pregnancy. BJOG. 2022 Jan;129(1):172. doi: 10.1111/1471-0528.16918. Epub 2021 Sep 29. No abstract available. PMID 34590410
- [Background] Kolding L, Ehrenstein V, Pedersen L, Sandager P, Petersen OB, Uldbjerg N, Pedersen LH. Antidepressant use in pregnancy and severe cardiac malformations: Danish register-based study. BJOG. 2021 Nov;128(12):1949-1957. doi: 10.1111/1471-0528.16772. Epub 2021 Jun 22. PMID 34036715
- [Background] Wolgast E, Lindh-Astrand L, Lilliecreutz C. Women's perceptions of medication use during pregnancy and breastfeeding-A Swedish cross-sectional questionnaire study. Acta Obstet Gynecol Scand. 2019 Jul;98(7):856-864. doi: 10.1111/aogs.13570. Epub 2019 Mar 20. PMID 30739330
- [Background] Bull FC, Al-Ansari SS, Biddle S, Borodulin K, Buman MP, Cardon G, Carty C, Chaput JP, Chastin S, Chou R, Dempsey PC, DiPietro L, Ekelund U, Firth J, Friedenreich CM, Garcia L, Gichu M, Jago R, Katzmarzyk PT, Lambert E, Leitzmann M, Milton K, Ortega FB, Ranasinghe C, Stamatakis E, Tiedemann A, Troiano RP, van der Ploeg HP, Wari V, Willumsen JF. World Health Organization 2020 guidelines on physical activity and sedentary behaviour. Br J Sports Med. 2020 Dec;54(24):1451-1462. doi: 10.1136/bjsports-2020-102955. PMID 33239350
- [Background] Reichetzeder C. Overweight and obesity in pregnancy: their impact on epigenetics. Eur J Clin Nutr. 2021 Dec;75(12):1710-1722. doi: 10.1038/s41430-021-00905-6. Epub 2021 Jul 6. PMID 34230629
- [Background] Goldstein RF, Abell SK, Ranasinha S, Misso M, Boyle JA, Black MH, Li N, Hu G, Corrado F, Rode L, Kim YJ, Haugen M, Song WO, Kim MH, Bogaerts A, Devlieger R, Chung JH, Teede HJ. Association of Gestational Weight Gain With Maternal and Infant Outcomes: A Systematic Review and Meta-analysis. JAMA. 2017 Jun 6;317(21):2207-2225. doi: 10.1001/jama.2017.3635. PMID 28586887
- [Background] Amezcua-Prieto C, Olmedo-Requena R, Jimenez-Mejias E, Hurtado-Sanchez F, Mozas-Moreno J, Lardelli-Claret P, Jimenez-Moleon JJ. Changes in leisure time physical activity during pregnancy compared to the prior year. Matern Child Health J. 2013 May;17(4):632-8. doi: 10.1007/s10995-012-1038-3. PMID 22569946
- [Background] Ribeiro MM, Andrade A, Nunes I. Physical exercise in pregnancy: benefits, risks and prescription. J Perinat Med. 2021 Sep 6;50(1):4-17. doi: 10.1515/jpm-2021-0315. Print 2022 Jan 27. PMID 34478617
- [Background] Sanchez-Polan M, Franco E, Silva-Jose C, Gil-Ares J, Perez-Tejero J, Barakat R, Refoyo I. Exercise During Pregnancy and Prenatal Depression: A Systematic Review and Meta-Analysis. Front Physiol. 2021 Jun 28;12:640024. doi: 10.3389/fphys.2021.640024. eCollection 2021. PMID 34262468
- [Background] Sanchez-Polan M, Silva-Jose C, Franco E, Nagpal TS, Gil-Ares J, Lili Q, Barakat R, Refoyo I. Prenatal Anxiety and Exercise. Systematic Review and Meta-Analysis. J Clin Med. 2021 Nov 24;10(23):5501. doi: 10.3390/jcm10235501. PMID 34884202
- [Background] Barakat R, Pelaez M, Cordero Y, Perales M, Lopez C, Coteron J, Mottola MF. Exercise during pregnancy protects against hypertension and macrosomia: randomized clinical trial. Am J Obstet Gynecol. 2016 May;214(5):649.e1-8. doi: 10.1016/j.ajog.2015.11.039. Epub 2015 Dec 15. PMID 26704894
- [Background] Monk C, Fifer WP, Myers MM, Sloan RP, Trien L, Hurtado A. Maternal stress responses and anxiety during pregnancy: effects on fetal heart rate. Dev Psychobiol. 2000 Jan;36(1):67-77. PMID 10607362
- [Background] Barakat R. An exercise program throughout pregnancy: Barakat model. Birth Defects Res. 2021 Feb 1;113(3):218-226. doi: 10.1002/bdr2.1747. Epub 2020 Jul 2. PMID 32613735